CLINICAL TRIAL: NCT01769508
Title: A Phase II Study With Lead-in Safety Cohort of 5-Fluorouracil, Oxaliplatin and Lapatinib in Combination With Radiation Therapy as Neoadjuvant Treatment for Patients With Localized HER2 Positive Esophagogastric Adenocarcinomas
Brief Title: Study of 5-FU, Oxaliplatin, & Lapatinib Combined With Radiation Therapy to Treat HER2 Positive Esophagogastric Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed due to slow accrual.
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 166
Record Dates: First submitted 2013-01-11; First posted 2013-01-16 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-05

CONDITIONS: HER2 Positive Esophagogastric Cancer
Keywords: Esophagogastric Adenocarcinoma; 5-Fluorouracil; Oxaliplatin; Lapatinib; Radiation Therapy; Surgery
MeSH Terms: interventions — Fluorouracil; Combined Modality Therapy; Oxaliplatin; Lapatinib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combined Therapy (Experimental): Combined Modality Treatment of Radiation therapy, 5-Fluorouracil, Oxaliplatin and Lapatinib followed by Surgery
  Interventions: Drug: 5-Fluorouracil; Drug: Oxaliplatin; Drug: Lapatinib; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: 5-Fluorouracil — 5-FU, 225 mg/m2 IVCI, during XRT.
  Other Names: Combined Modality Treatment
Drug: Oxaliplatin — Oxaliplatin, 85 mg/m2 IV, Days 1, 15, 29.
  Other Names: Combined Modality Treatment
Drug: Lapatinib — Lapatinib, Continuous PO daily dosing during XRT, dose determined during lead in portion
  Other Names: Combined Modality Treatment
Radiation: Radiation Therapy — Radiation therapy, 50.4 Gy (1.8 Gy/day or 28 fractions) M-F, Weeks1-6

SUMMARY:
With improvements in response rate and survival seen for HER2 positive patients treated with HER2 blockade in the metastatic setting, the use of HER2 blockade in the neoadjuvant setting to increase antitumor effect shows promise. Patients with previously untreated localized HER2 positive esophageal, GE junction and gastric adenocarcinomas will be enrolled. Patients meeting all inclusion/exclusion criteria will receive neoadjuvant treatment with concurrent chemotherapy and radiation therapy beginning on day 1 of treatment. During the lead-in safety portion, the optimal dose of lapatinib will be determined.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, Phase II study with a lead-in safety cohort. The study will evaluate the combination of 5-Fluorouracil, Oxaliplatin and Lapatinib with radiation therapy as neoadjuvant treatment for patients with previously untreated localized HER2 positive esophagogastric adenocarcinomas. Approximately 12 patients will be enrolled in the lead-in cohort to evaluate the safety of the combination. Following the lead-in cohort, Phase II will commence and up to 30 additional patients may be treated. The starting doses will be administered as follows:

5-FU 225 mg/mg2 continuous intravenous (IV) infusion Days 1 - 42 during XRT; Oxaliplatin 85 mg/m2 Days 1, 15 and 29, given by IV infusion, per institutional standard; Lapatinib Continuous PO daily dosing during XRT (final dose determined during lead-in cohort).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Stage I, II, or III adenocarcinoma of the esophagus (lower ⅓), GE junction, or gastric cardia.
* Clinical stage I, II, or III as assessed by required baseline staging. In addition, patients with celiac node involvement (stage IVa) are eligible.
* Patients must be surgical candidates based on stage and location of disease as well as other medical conditions and risk factors.
* Positive HER2 status (overexpression and/or amplification of HER2 in primary tumor) as defined by FISH (HER2 FISH positivity).
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 or 1.
* Patient must be able to swallow and absorb oral medication.
* Patients must have an indwelling central venous access catheter.
* Adequate hematologic, renal, and hepatic function:
* Known brain or leptomeningeal metastases.
* Male patients willing to use adequate contraceptive measures.
* Female patients who are not of child-bearing potential, and female patients of child-bearing potential who agree to use adequate contraceptive measures, who are not breastfeeding, and who have a negative serum or urine pregnancy test within 72 hours prior to start of treatment.
* Life expectancy ≥ 12 weeks.
* Age ≥18 years of age.
* Willingness and ability to comply with trial and follow-up procedures.
* Ability to understand the nature of this trial and give written informed consent.

Exclusion Criteria:

* Patients with evidence of distant metastases are ineligible, as are patients who are not potential surgical candidates based on location or extent of local disease. Patients with celiac nodal disease (Stage IVa) will be allowed on study.
* Previous anti-cancer treatment for esophageal, GE junction, or gastric cancer.
* Any other investigational agents within the 28 days prior to day 1 of the study.
* Known active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).
* Concurrent treatment with drugs known to be strong inhibitors or inducers of isoenzyme CYP3A that cannot be discontinued or switched to different medication prior to starting study drug.
* Concurrent use of St. John's wort and grapefruit /grapefruit juice ≤7 days prior to starting study drug is not allowed.
* Ongoing treatment with full-dose warfarin or its equivalent. Prophylactic treatment with 1 mg daily of warfarin and/or low molecular weight heparin is allowed.
* History of any other disease, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of a novel regimen, or that might affect interpretation of the results of this study or render the subject at high-risk for treatment complications.
* Active gastrointestinal (GI) disease or other condition that in the opinion of the investigator will interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy (e.g. ulcerative disease, uncontrolled nausea, or vomiting).
* Poorly controlled or clinically significant atherosclerotic vascular disease
* A serious active infection at the time of treatment, or another serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
* Known diagnosis of human immunodeficiency virus (HIV), Hepatitis B (HBV) or Hepatitis C (HCV).
* Presence of other active cancers, or history of treatment for invasive cancer ≤5 years. Patients with stage I cancer who have received definitive local treatment at least 3 years previously, and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (i.e. non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Inability or unwillingness to comply with study and/or follow-up procedures outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johanna C Bendell, MD, Study Chair — SCRI Development Innovations, LLC
Locations (9):
- United States (9):
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Woodlands Medical Specialists, Pensacola, Florida
  - Florida Cancer Specialists-North, St. Petersburg, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Grand Rapids Oncology Program, Grand Rapids, Michigan
  - Oncology Hematology Care, Cincinnati, Ohio
  - Chattanooga Oncology and Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee

REFERENCES:
- [Derived] Shepard G, Arrowsmith ER, Murphy P, Barton JH Jr, Peyton JD, Mainwaring M, Blakely L, Maun NA, Bendell JC. A Phase II Study with Lead-In Safety Cohort of 5-Fluorouracil, Oxaliplatin, and Lapatinib in Combination with Radiation Therapy as Neoadjuvant Treatment for Patients with Localized HER2-Positive Esophagogastric Adenocarcinomas. Oncologist. 2017 Oct;22(10):1152-e98. doi: 10.1634/theoncologist.2017-0186. Epub 2017 Aug 1. PMID 28765502

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combined Therapy
Started | 12
Completed | 6
Not Completed | 6
Not completed — Death | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: All enrolled and treated patients
Arm/Group | Combined Therapy
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 64 [42 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate (pCR Rate)
Description: Defined as the absence of invasive tumor in esophagogastric and lymph node tissue removed at time of surgery, as judged by the local pathologist. An improvement in pCR rate from 30 percent (historical) to 50 percent is the primary efficacy endpoint.
Time Frame: 18 months
Population: All patients who underwent surgery
Measure: Number; unit: participants
Arm/Group | Combined Therapy
Number analyzed (Participants) | 3
participants | 1

2. Primary Outcome: Safety and Optimal Dose of Regimen
Description: An additional primary objective is to evaluate the safety and optimal dose of lapatinib when added to 5-FU, oxaliplatin and radiation therapy.
Time Frame: 18 months
Measure: Number; unit: mg QD Lapatinib
Arm/Group | Combined Therapy
Number analyzed (Participants) | 12
mg QD Lapatinib | 750

3. Secondary Outcome: Progression Free Survival (PFS)
Description: The Percentage of Patients Who Experience an Objective Benefit From Treatment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combined Therapy
Number analyzed (Participants) | 12
months | 3.253 [1.183 to 6.768]

4. Secondary Outcome: Toxicity Profile for Treated Patients
Description: Defined as the frequency of adverse events for patients who received at least one dose of study treatment, and assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0.
Time Frame: 18 months
Population: All treated patients
Measure: Number; unit: participants
Arm/Group | Combined Therapy
Number analyzed (Participants) | 12
participants
  Nausea | 9
  Diarrhea | 7
  Fatigue | 6
  Vomiting | 5
  Mucositis | 4
  Stomatitis | 3
  Anemia | 2
  Anorexia | 2
  Constipation | 2
  Dehydration | 2
  Dysesthesia | 2
  Dysgeusia | 2
  Dysphagia | 2
  Esophagitis | 2
  Cold sensitivity | 2
  Hypokalemia | 2
  Peripheral sensory neuropathy | 2
  Thrombocytopenia | 2
  Rash | 2
  Thromboembolic event | 2

5. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression is defined as the time between day 1 cycle 1 and time to first documented disease progression. Disease progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combined Therapy
Number analyzed (Participants) | 12
months | 6.768 [6.604 to 6.965]

6. Secondary Outcome: Overall Survival (OS)
Description: The Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combined Therapy
Number analyzed (Participants) | 12
months | NA [NA to NA] — Median OS has not been reached as not enough death events have occurred at this time point

ADVERSE EVENTS:
Time Frame: 26 months
Arm/Group | Combined Therapy
Serious Adverse Events (participants affected / at risk) | 6/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Therapy (N=12)
Allergic Reaction (Immune system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Death NOS (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Eye disorders - Other, vision changes (Eye disorders) | 1
General disorders and administration site conditions - Other, hemorrhage (General disorders) | 1
Heart Failure (Cardiac disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Infections and infestations - Other, pneumonia (Infections and infestations) | 1
Metabolism and nutrition disorders - Other, malnutrition (Metabolism and nutrition disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, benign pituitary tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Therapy (N=12)
Nausea (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 6
Vomiting (Gastrointestinal disorders) | 5
Mucositis (Gastrointestinal disorders) | 4
Weight Loss (Investigations) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Dysphagia (Gastrointestinal disorders) | 3
Gastrointestinal Disorders - Other, Stomatitis (Gastrointestinal disorders) | 3
Anemia (Blood and lymphatic system disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Dysesthesia (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Esophagitis (Gastrointestinal disorders) | 2
General Disorders And Administration Site Conditions - Other, Cold Sensitivity (General disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 2
Platelet Count Decreased (Investigations) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Thromboembolic Event (Vascular disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Allergic Reaction (Immune system disorders) | 1
Cardiac Arrest (Cardiac disorders) | 1
Death Nos (General disorders) | 1
Edema Limbs (General disorders) | 1
Eye Disorders - Other, Vision Changes (Eye disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
General Disorders And Administration Site Conditions - Other, Hemorrhage (General disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Infections And Infestations - Other, Pneumonia (Infections and infestations) | 1
Insomnia (Psychiatric disorders) | 1
Metabolism And Nutrition Disorders - Other, Malnutrition (Metabolism and nutrition disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps) - Other, Pituitary Macroadenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Paresthesia (Nervous system disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Skin Infection (Infections and infestations) | 1
White Blood Cell Decreased (Investigations) | 1

LIMITATIONS AND CAVEATS:
Trial closed early due to slow accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites